CLINICAL TRIAL: NCT00695877
Title: A Phase I Randomized, Double-blind, Placebo Controlled Dose Escalation Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Adenovirus Serotype 5 HVR48 HIV-1 Vaccine (Ad5HVR48.ENVA.01) in Healthy, HIV-1 Uninfected Adults (Ad5HVR48.ENVA.01 (rAd5HVR48) HIV-1/IPCAVD-002 Vaccine Study)
Brief Title: Safety and Immune Response to a Recombinant Adenovirus HIV-1 Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ad5HVR48.ENVA.01/IPCAVD-002; 10701 (Registry Identifier: DAIDS ES Registry Number); Ad5HVR48.ENVA.01/ IPCAVD-002
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 3 injections of rAd5.ENVA.48 HIV-1 vaccine or placebo at 1 x 10^9 virus particles (VP) given at Days 0, 28, and 168
  Interventions: Biological: Ad5.ENVA.48 HIV-1 vaccine
- 2 (Experimental): 3 injections of rAd5.ENVA.48 HIV-1 vaccine or placebo at 1 x 10^10 virus particles (VP) given at Days 0, 28, and 168
  Interventions: Biological: Ad5.ENVA.48 HIV-1 vaccine
- 3 (Experimental): 3 injections of rAd5.ENVA.48 HIV-1 vaccine or placebo at 1 x 10^11 virus particles (VP) given at Days 0, 28, and 168
  Interventions: Biological: Ad5.ENVA.48 HIV-1 vaccine
- 4 (Experimental): 1 injection of rAd5.ENVA.48 HIV-1 vaccine or placebo at a dose determined by the safety data from Arms 1, 2 and 3 given at Day 0.
  Interventions: Biological: Ad5.ENVA.48 HIV-1 vaccine

INTERVENTIONS:
Biological: Ad5.ENVA.48 HIV-1 vaccine — Recombinant adenovirus serotype 5 HIV-1 vaccine

SUMMARY:
Successful control of the HIV epidemic will require a safe and effective vaccine to be developed. A successful vaccine will need to stimulate a widespread immune response. The purpose of this study is to determine the safety of and immune response to an adenovirus serotype HIV vaccine in HIV uninfected adults.

DETAILED DESCRIPTION:
Control of the HIV pandemic can only be achieved with the development of a safe and effective preventive HIV vaccine. A vaccine that will prevent HIV infection will elicit a strong immune response from both CD4 and CD8 cells. Recombinant adenovirus serotype vectors have been shown to elicit just such a response. The purpose of this study is to determine the safety and immunogenicity of the recombinant adenovirus serotype 5 preventive HIV-1 vaccine.

This study will last 18 to 24 months. Participants will be randomly assigned to one of four arms that will receive vaccine or placebo administered via intramuscular injection. Participants in Arms 1, 2, and 3 will all receive 3 injections. Participants in Arm 4 will receive one injection. For most participants, there will be 10 study visits in this study; for participants in Arm 4, there will be only 7 visits. For Arms 1, 2, and 3, study visits will occur at baseline and on Days 0, 14, 28, 42, 56, 168, 182,196, and 365. Participants in Arms 1, 2, and 3 will receive injections on Days 0, 28, and 168. For participants in Arm 4, study visits will occur at baseline and on Days 0, 14, 28, 56, 168 and 365. Participants in Arm 4 will receive one injection only, on Day 0. Participants will be asked to record their temperature and other side effects in a symptom log for 3 days after each injection. Risk reduction/pregnancy prevention counseling and physical exams will occur at all visits. At most visits, blood, urine, and oral swab collection will occur. Samples collected will be stored for future testing. HIV testing and pregnancy testing will occur at select visits. At Years 2, 3, 4, and 5, participants will be followed-up by telephone, e-mail, or study visit to collect vital status, and information about any development of significant disability or incapacity, hospitalizations, or congenital anomalies. At these follow-up visits, blood collection will be optional.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Normal hematological, hepatic and renal functions
* Demonstrated understanding of study
* Willing to receive HIV test results
* HIV-1 and -2 uninfected
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (anti-HCV) negative antibody or negative HCV PCR if anti-HCV is positive
* Adequate contraception. For more information on this criterion can be found in the protocol.

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first injection. Participants taking corticosteroid nasal spray or topical corticosteroids are not excluded.
* Blood products within 120 days prior to first injection
* Immunoglobulin within 60 days prior to first injection
* Investigational agents within 30 days prior to first injections
* Live attenuated vaccine within 30 days prior to first injection
* Any vaccine that is not a live attenuated vaccine within 14 days prior to first injection
* Any clinically significant medical condition that, in the opinion of the investigator, may interfere with the study
* Any medical, psychiatric, occupational, or social condition or responsibility that, in the opinion of the investigator, would interfere with the study
* Serious adverse reaction to vaccines. Participants who had a nonanaphylactic adverse reaction to pertussis vaccine as a child are not excluded.
* Known autoimmune disease
* Known immunodeficiency
* Asthma other than mild, well-controlled asthma
* Diabetes mellitus type 1 or 2
* Thyroidectomy or thyroid disease in the12 months prior to study entry
* Angioedema in the 3 years prior to study entry
* Hypertension. More information on this criterion can be found in the protocol.
* Body mass index (BMI) of 40 or higher OR BMI of 35 or greater, if other cardiovascular risk factors. More information on this criterion can be found in the protocol.
* Bleeding disorder
* Malignancy, unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder or occurrence of seizure in the 3 years prior to study entry. Participants who have not required medications or had a seizure for prior 3 years are not excluded.
* Absence of spleen
* Individuals at high-risk of acquiring HIV infection
* Presence of pre-existing neutralizing antibodies for Adenovirus 5 or 48
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-02-08 (Actual); Primary Completion 2012-12-11 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Local and systemic adverse reactions | Throughout study

SECONDARY OUTCOMES:
Humoral Immune response | Throughout study
Cell mediated immunity | Throughout study
Genotyping | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Study Chair — Brigham and Women's Hospital; Dan Barouch, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Brigham and Women's Hosp. Novel Adenoviral Vector Prophylactic HIV Vaccine Non-Network CRS, Boston, Massachusetts, United States

REFERENCES:
- [Background] Priddy FH, Brown D, Kublin J, Monahan K, Wright DP, Lalezari J, Santiago S, Marmor M, Lally M, Novak RM, Brown SJ, Kulkarni P, Dubey SA, Kierstead LS, Casimiro DR, Mogg R, DiNubile MJ, Shiver JW, Leavitt RY, Robertson MN, Mehrotra DV, Quirk E; Merck V520-016 Study Group. Safety and immunogenicity of a replication-incompetent adenovirus type 5 HIV-1 clade B gag/pol/nef vaccine in healthy adults. Clin Infect Dis. 2008 Jun 1;46(11):1769-81. doi: 10.1086/587993. PMID 18433307
- [Background] Stevens W, Kamali A, Karita E, Anzala O, Sanders EJ, Jaoko W, Kaleebu P, Mulenga J, Dally L, Fast P, Gilmour J, Farah B, Birungi J, Hughes P, Manigart O, Stevens G, Yates S, Thomson H, von Lieven A, Krebs M, Price MA, Stoll-Johnson L, Ketter N. Baseline morbidity in 2,990 adult African volunteers recruited to characterize laboratory reference intervals for future HIV vaccine clinical trials. PLoS One. 2008 Apr 30;3(4):e2043. doi: 10.1371/journal.pone.0002043. PMID 18446196
- [Derived] Baden LR, Walsh SR, Seaman MS, Johnson JA, Tucker RP, Kleinjan JA, Gothing JA, Engelson BA, Carey BR, Oza A, Bajimaya S, Peter L, Bleckwehl C, Abbink P, Pau MG, Weijtens M, Kunchai M, Swann EM, Wolff M, Dolin R, Barouch DH. First-in-human evaluation of a hexon chimeric adenovirus vector expressing HIV-1 Env (IPCAVD 002). J Infect Dis. 2014 Oct 1;210(7):1052-61. doi: 10.1093/infdis/jiu217. Epub 2014 Apr 8. PMID 24719474